CLINICAL TRIAL: NCT00529815
Title: A Pilot Study to Determine the Impact of Real-Time Continuous Glucose Monitoring (CGM) on Patients With Type 2 Diabetes
Brief Title: Continuous Glucose Monitoring in Patients With Type 2 Diabetes
Acronym: CGM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Col. Robert A. Vigersky MC, MD, WRAMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WU # 07-13023
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Continuous; blood; glucose; monitoring; diabetes; type2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1CGM and SBGM (Experimental): Intervention group will alternate the use of the CGM with episodic self blood glucose monitoring for four cycles of two weeks using the CGM and episodic SBGM and one week only using episodic SBGM during the 12 week study.
  Interventions: Device: Continuous Glucose Monitor
- 2 SBGM (Active Comparator): The control group (SBGM) will be instructed in the use of the Accuchek Aviva glucometer.
  Interventions: Device: Glucometer

INTERVENTIONS:
Device: Continuous Glucose Monitor — The intervention group will alternate the use of the CGM with episodic self blood glucose monitoring for four cycles of two weeks using the CGM and episodic SBGM and one week only using episodic SBGM during the 12 week study.
  Arms: 1CGM and SBGM
Device: Glucometer — The control group (SBGM) will be instructed in the use of the Accuchek Aviva glucometer.
  Arms: 2 SBGM

SUMMARY:
The purpose of this pilot study is to determine if a Real-Time Continuous Glucose Monitoring System (CGMS) is a more effective method of improving glycemic control in patients with type 2 diabetes than is episodic self blood glucose monitoring(SBGM) in the both the short- and long-term. CGMS, which includes a sensor that can be self- inserted under the skin and a discrete monitor that records and displays blood sugar levels nearly continuously, allows for real time blood glucose monitoring. This will be a prospective, randomized control trial comparing participants with type II diabetes use of CGMS versus SBGM. The primary endpoint will be improvement of glycemic control as measured by glycosylated hemoglobin (A1C). The secondary endpoints will compare mean daily glucose levels, the number of both hypoglycemic and hyperglycemic events, the amount of time spent in target blood glucose, and the perceived level of diabetes-related stress between the two groups. Participants will be randomized to either the control (SBGM) or intervention (CGMS) group. Subjects in the intervention group will alternate the use of the CGMS with episodic self blood glucose monitoring for four cycles of two weeks during the 12 week study. The control group will perform episodic SBGM throughout the study. The intensified monitoring schedules for both groups will end at the end of week 12, but glycemic control measurement by A1C will continue through 52 weeks. A1C levels will be drawn at 0, 12, 24, 38, and 52 weeks. Mean daily blood glucose levels, number of hypo and hyperglycemic events, and duration of time spent in target blood glucose range will be downloaded from patients' meters periodically throughout the study. The SF-8, a general quality of life questionnaire for people with chronic disease, and Problem Areas in Diabetes (PAID), a diabetes-related quality of life questionnaire, will be completed at the beginning and end of the study. The results of this study may help highlight which blood glucose monitoring methods are most likely to improve patients' ability to achieve and maintain target levels of glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Known Type 2 diabetes for at least 3 months
3. Diet controlled, on oral therapy, on basal insulin (e.g. glargine), or on oral therapy and a basal insulin
4. A1C levels between 7% and 12%.
5. Able to independently measure and read finger stick blood glucose levels with the Accu-chek Aviva glucometer and the DexCom Continuous Glucose Monitoring device (DexCom DTS-7).
6. Subjects will have attended a American Diabetes Association recognized Diabetes Self-Management Education (DSME) program at one of the WRHCS military treatment facilities (MTFs) within the past five years.
7. Willing to avoid or minimize use of acetaminophen (Tylenol) and all acetaminophen- containing products such as most over-the-counter (OTC) medications during the study period (Appendix 5)..

Exclusion Criteria:

1. Female subjects who are pregnant, lactating, planning to become pregnant, or without a safe contraceptive method.
2. A1C levels are less than 7 or greater than 12.
3. Subjects who are taking glucocorticoids, amphetamines, anabolic, or weight-reducing agents during the course of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
This study will determine if a real-time continuous glucose monitoring system is a more effective method of improving glycemic control in patients with type 2 diabetes than is episodic self blood glucose monitoring in the both the short- and long-term. | March 1, 2010

SECONDARY OUTCOMES:
The results of this study could also provide information on the impact of the two methods of glycemic monitoring on number of hypoglycemic and hyperglycemic events, and quality of life. | March 1, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Vigersky, MD, Principal Investigator — WRAMC
Locations (1):
- Walter Reed Army Hospital Center, Washington D.C., District of Columbia, United States